CLINICAL TRIAL: NCT01260675
Title: A Study to Assess the Pharmacokinetic Profile of an Investigational Formulation of Buprenorphine HCl/Naloxone HCl 8mg/2mg Capsules Relative to the Pharmacokinetic Profile of Suboxone® (Buprenorphine HCl/Naloxone HCl 8mg/2mg Sublingual Tablets).
Brief Title: Study to Assess the PK Profile of NanoBUP Capsules Relative to Suboxone
Status: Completed | Type: Observational
Sponsor: NanoSHIFT LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009-BUP-NT/002
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: phase 1 study; volunteers
MeSH Terms: interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NanoBUP Capsules: Investigational Formulation of Buprenorphine HCl/Naloxone HCl 8 mg/2 mg oral capsules
  Interventions: Drug: Buprenorphine HCl/Naloxone HCl
- Suboxone Sublingual Tablets: Buprenorphine HCl/Naloxone HCl 8 mg/2 mg sublingual tablets
  Interventions: Drug: Buprenorphine HCl/Naloxone HCl

INTERVENTIONS:
Drug: Buprenorphine HCl/Naloxone HCl
  Other Names: Suboxone

SUMMARY:
Phase 1 study to determine the pharmacokinetic profile of NanoBUP Capsules to Suboxone.

DETAILED DESCRIPTION:
The pharmacokinetics of an orally administered investigational buprenorphine hydrochloride/naloxone hydrochloride 2 mg/0.5 mg capsule formulation will be studied. This is a single-dose, two period, two treatment, crossover comparative bioavailability study under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breastfeeding female.
* Subject must be between 18 and 55 years of age (inclusive).
* Subject's Body Mass Index (BMI) must be between 18 and 30 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Female subjects - not surgically sterile for at least 6 months or at least 2 years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, hormonal (oral, implant, transdermal, vaginal, or injection) in use at least 3 consecutive months prior to the first dose of study medication, double barrier (condom with spermicide; diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to start of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of the confinement period and return for any outpatient visits

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, metabolic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* A clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening.
* History or presence of allergic or adverse response to buprenorphine, naloxone, naltrexone, opioids, or any comparable or similar products.
* Been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Donated blood or plasma within 30 days prior to the first dose of study medication.
* Participated in another clinical trial within 30 days prior to the first dose of study medication.
* Used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs, such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Smoked or used tobacco products within 60 days prior to the first dose of study medication.
* History of substance abuse or dependence (including alcohol, opioids, or intravenous drug abuse)
* Is a female with a positive pregnancy test result.
* A positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* A positive urine alcohol test at screening or a positive ethanol breath test at check-in for the study period or has consumed alcohol within 48 hours prior to screening or check-in for the study period.
* Had a positive test for, or has been treated for hepatitis B, hepatitis C, or HIV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01-31 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of NanoBUP Capsules relative to Suboxone | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Natalino, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States